CLINICAL TRIAL: NCT04327674
Title: The Use of Focused Lung Ultrasound in Patients Suspected of COVID-19
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-FLUS
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID is a major health problem causing massive capacity problems at hospitals. Rapid and accurate diagnostic workflow is of paramount importance. Access to radiological diagnostics tools such as x-ray or computed tomography of the chest are limited even in high-resource settings.

Focused lung ultrasound, FLUS, is a point-of-care diagnostic tool that allows rapid and on-site assessment of lung abnormalities. No transportation of the patient is required thus lowering risk of spreading SAR-CoV- inside the hospital.

This study aims to explore the diagnostic value of FLUS in the COVID-19 pandemic and to explore if FLUS findings can predict risk of respiratory failure.

DETAILED DESCRIPTION:
COVID-19 is defined as an infectious disease caused by SAR-CoV-2 virus. It results in pneumonia and sometimes respiratory failure. SARS-CoV-2 pandemic has led to massive strain on health care facilities. A large proportion of the population is at risk of COVID-19 and some estimates suggest that up to 15% will need hospitalization. Such number of patients strains the health care system to its maximum as capacity has limitations even in highly developed countries.

Early reports estimate that more than 80% of patients admitted to hospital with COVID-19 have abnormal findings on chest radiographs1. Thus, imaging seems to be an important part of the diagnostic work-up. In most hospitals however, access to CT-scanning of the thorax of all patients with COVID-19 or with suspicion of CODIV-19 is unrealistic due to restricted capacity. Chest radiographs are faster and easier to do, but may require transportation of the patient to the department of radiology which carries a risk of virus spreading in the hospital. On-site chest radiograph is often of such low quality that diagnosis or follow-up will be difficult.

Focused ultrasound examination of the lungs, FLUS, is a diagnostic tool that can show changes in the lung parenchyma due to pneumonia. FLUS is a bed-side examination performed by the physician which results in reduced risk of in-hospital virus contamination. Furthermore, results from FLUS are immediately available to the physician. This allows rapid decision-making which is essential in cases of high patient burdens as seen in the COVID-19 pandemic.

Furthermore, SARS-CoV-2 positive patients with pneumonia may be at higher risk of respiratory failure than those without pneumonia. Identifying patients at high risk can qualify decisions about monitoring level and organization of intensive care resources. Conversely, patient with COVID-19 symptoms but without pneumonic FLUS finding could likely be managed as out-patients. Such a risk-stratification may optimize the allocation of limited healthcare resources and reserve in-hospital capacity to those patients who needs it.

Hypothesis:

FLUS can risk-stratify patients with COVID-19 symptoms. FLUS can predict respiratory failure in patients with COVID-19 pneumonia. FLUS can diagnose COVID-19 pneumonia with high sensitivity and specificity using PCR-test and chest radiograph as reference.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of COVID-19 requiring contact to a hospital.

Exclusion Criteria:

* Age less than 18 years
* Previous enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who have symptoms on COVID-19 and is seen at a hospital.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2020-03-14 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren H Skaarup, Principal Investigator — Aarhus Universitets Hospital
Locations (2):
- Denmark (2):
  - Lungemedicinsk Forskningsafdeling. Aarhus University Hospital, Aarhus
  - Regionshospitalet Horsens., Horsens

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Focused Lung Ultrasound: All patients admitted to hospital with symptoms of COVID-19 or PCR confirmed SARS-CoV-2 infection.
Period: Overall Study
Arm/Group | Focused Lung Ultrasound
Started | 417
Completed | 398
Not Completed | 19
Not completed — Protocol Violation | 19

BASELINE CHARACTERISTICS:
Groups:
- FLUS: All patients admitted to hospital with symptoms of COVID-19 or PCR confirmed SARS-CoV-2 infection
Arm/Group | FLUS
Number analyzed (Participants) | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189
  Male | 209
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 398

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Ventilation
Description: Number of patients on mechanical ventilation.
Time Frame: During admission, an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | FLUS
Number analyzed (Participants) | 398
Participants | 21

2. Secondary Outcome: FLUS Findings and Admission to Intensive Care.
Description: Intensive care admissions
Time Frame: During admission, an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | FLUS
Number analyzed (Participants) | 398
Participants | 28

3. Secondary Outcome: SAR-CoV-2 PCR-test Result.
Description: Positive SAR-CoV-2 PCR-test
Time Frame: During admission, an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | FLUS
Number analyzed (Participants) | 398
Participants | 227

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | FLUS
All-Cause Mortality (participants affected / at risk) | 47/398
Serious Adverse Events (participants affected / at risk) | 398/398
Other Adverse Events (participants affected / at risk) | 0/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLUS (N=398)
Admission to hospital (Respiratory, thoracic and mediastinal disorders) | 398 (398)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04327674/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04327674/SAP_001.pdf